CLINICAL TRIAL: NCT06965816
Title: Using Neuroimaging to Early Diagnose Alzheimer's Disease Through Hippocampal Atrophy Assessment
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0030_IMAGERIE
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer's Disease; Hippocampus; Brain Atrophy; Magnetic Resonance Imaging; Leukoaraiosis; Neurodegenerative Diseases; Cortical and Subcortical Atrophy
MeSH Terms: conditions — Leukoaraiosis; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alzheimer Group: Alzheimer's patients
- Control Group: Unreached witnesses

SUMMARY:
This study aims to better understand Alzheimer's disease by looking at brain scans, specifically MRI images, to detect early signs of brain changes linked to the disease. Researchers are focusing on the hippocampus, a part of the brain that shrinks in people with Alzheimer's. The study will also explore other brain changes that often happen alongside hippocampal shrinkage. By analyzing these brain images, the study hopes to find ways to diagnose Alzheimer's earlier and more accurately using advanced imaging techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a brain MRI (3D T1 Bravo and Cube FLAIR sequences) between January 2018 and June 2022.
* Diagnosis of Alzheimer's disease (for the Alzheimer group).
* No neurological disease for control group participants.
* Complete clinical and biological assessments available.
* Quality imaging without motion artifacts.

Exclusion Criteria:

* Incomplete clinical or radiological data.
* Poor image quality (e.g., motion artifacts).
* Presence of other neurodegenerative or psychiatric disorders.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be selected from a retrospective cohort of patients who underwent brain MRI scans (3D T1 Bravo and Cube FLAIR sequences) between January 2018 and June 2022. The study population includes two groups: patients diagnosed with Alzheimer's disease based on clinical and biological assessments, and cognitively healthy individuals with no history of neurological or psychiatric disorders, serving as controls.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Hippocampal Volume Measured by 3D MRI | Retrospective analysis between January 2018 and June 2022
  Objective volumetric measurement of the right and left hippocampus using 3D T1 Bravo MRI sequences, allowing quantification of hippocampal atrophy.

CONTACTS AND LOCATIONS:
Locations (1):
- France, Saint-Denis, France

IPD SHARING:
Plan to Share IPD: No